CLINICAL TRIAL: NCT02112188
Title: Adaptation of Individual Meaning-Centered Psychotherapy for Chinese Immigrant Cancer
Brief Title: Meaning-Centered Counseling for Chinese Patients Who Are Being Treated for Advanced Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Queens Cancer Center of Queens Hospital (Other); Charles B. Wang Community Health Center (CBWCHC) (Unknown); American Cancer Society - Asian Initiatives (Other); New York Coalition for Asian American Mental Health (NYCAAMH) (Unknown); New York Hospital Queens (Other); Chinese Christian Herald Crusades (CCHC) (Other); Cheung and Kan Medical Group, PLLC (Unknown); The City College of New York (Other); MediSys Health Network (Other)
Responsible Party: Sponsor
Other Study IDs: 14-076
Record Dates: First submitted 2014-04-07; First posted 2014-04-11 (Estimated); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Advanced Cancer
MeSH Terms: interventions — Clinical Trials, Phase IV as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Chinese patients with advanced cancer: IMCP intervention to be culturally & linguistically tailored for Chinese cancer patients. This study will be carried out in 3 phases: 1) formative research & 2) adaptation. For this application we will continue the formative research (phase 1) by conducting 20 to 30 indepth interviews with Chinese immigrants with advanced cancer to inform the adaptation of the intervention. Results of the patient in-depth interviews will inform how to adapt the IMCP process & session themes to reflect the needs of the community. In the adaptation phase (phase 2) the Breitbart IMCP research team (including Drs. Breitbart, Lichtenthal, & Applebaum), Drs. Leng, Gany, & Ms. Huang will discuss a priori adaptations to the intervention. Potential changes to the process & content will be discussed. Adaptations will be incorporated in a modified IMCP-Ch treatment manual, therapist checklist/outline & Treatment Integrity Coding Manual. PHASE 3, 4 Conduct feasibility study of IMCP-Ch for Chinese cancer patients.
  Interventions: Behavioral: In-depth Patient Interviews; Behavioral: Adaptation of IMCP for Chinese Immigrant Cancer Patients; Behavioral: Individual Meaning-Centered Psychotherapy for Chinese (IMCP-Ch) (For Phase 3 and Phase 4)

INTERVENTIONS:
Behavioral: In-depth Patient Interviews
Behavioral: Adaptation of IMCP for Chinese Immigrant Cancer Patients
Behavioral: Individual Meaning-Centered Psychotherapy for Chinese (IMCP-Ch) (For Phase 3 and Phase 4) — The six sessions will be delivered every or every other week over a span of 6-16 weeks, depending on participant and interventionist availability. Sessions may also be delivered within 2 weeks to accommodate schedules. Sessions will take place via MSK-approved videoconferencing platforms (e.g. Zoom) or by telephone, depending on participant preference. The IMCP-Ch intervention will be delivered via telehealth in Mandarin Chinese by a bilingual interventionist or in English (for bilingual Chinese and English-speaking patients who prefer English) by an English-speaking therapist or through English-to-Mandarin Remote Simultaneous Medical Interpretation (RSMI), depending on participants' preference. All Phase 4 sessions will be digitally audio-recorded and saved to Zoom cloud. Cloud recording will be deleted from Zoom after the files have been uploaded.

SUMMARY:
The purpose of the study is to modify a type of counseling called "Individual Meaning Centered Psychotherapy" to meet the needs of Chinese cancer patients. Many cancer patients use counseling or other resources to help cope with the emotional burden of their illnesses. Counseling often helps them cope with cancer by giving them a place to express their feelings. "Meaning-Centered" counseling aims to teach cancer patients how to maintain or even increase a sense of meaning and purpose in their lives, despite cancer.

DETAILED DESCRIPTION:
Phases 1 and 2: Formative Research and Adaptation This is a study to adapt the IMCP intervention to be culturally and linguistically tailored for Chinese cancer patients. This study will be carried out in two phases: 1) formative research and 2) adaptation. Preliminary formative research has begun in our study exploring community needs and priorities through exemption application X13-034. For this application we will continue the formative research (phase 1) by conducting 12 in-depth interviews with Chinese immigrants with advanced cancer to inform the adaptation of the intervention. Results of the patient in-depth interviews will inform how to adapt the IMCP process and session themes to reflect the needs of the community. In the adaptation phase (phase 2) the Breitbart IMCP research team (including Drs. Breitbart, Lichtenthal, and Applebaum), Drs. Leng, Gany, and Ms. Huang will discuss a priori adaptations to the intervention. Potential changes to the process and content will be discussed. Adaptations will be incorporated in a modified IMCP-Ch treatment manual, therapist checklist/outline and Treatment Integrity Coding Manual.

Phase 3: Proof-of-concept" single-arm pilot trial of IMCP-Ch This phase will feature an open feasibility study using a pretest vs. posttest design, with the intervention to be delivered via telehealth in Mandarin Chinese by a bilingual interventionist or by an English-speaking therapist in English (for bilingual Chinese and English-speaking patients who prefer English) or through English-to-Mandarin Remote Simultaneous Medical Interpretation (RSMI), depending on participants' preference

Added a new phase (Phase 4), to examine the effects of using remote interpreting modalities to deliver IMCP-CH to Mandarin-speaking patients with advanced cancer; and (2) to add a minimum distress level for eligibility in order to align trial eligibility criteria with those employed in prior MCP trials, which used a DistressThermometer (DT) cutoff of >4 to identify patients with clinically significant distress (participants who do not meet this criteria will be enrolled in Phase 3). Phase 4 will employ a three-arm pilot randomized controlled trial (RCT) design to test the feasibility and acceptability of using (1) Remote Consecutive Medical Interpretation (RCMI), (2) Remote Simultaneous Medical Interpretation (RSMI) and (3) bilingual provider (control/gold standard) in delivering IMCP-Ch.

ELIGIBILITY:
Inclusion Criteria:

Phases 1 and 2:

Interview Inclusion Criteria (per self-report):

* Non-US born;
* Of Chinese descent;
* Age 21 years through 80 years;
* Language spoken: Mandarin and/or English
* Diagnosis of Stage IV cancer (any type).

Phase 3:

* Stage III or IV cancer (per self-report or on the MSKCC EMR). If traditional staging does not apply (i.e. for leukemia), we can allow patient deemed by provider to have poor prognosis/roughly equivalent to Stage III or IV to be referred.
* Age 18 or older
* Of Chinese descent
* Mandarin-speaking
* Have an estimated life expectancy of at least 6 months (per self-report or on the MSKCC EMR)
* Resides in New York State or New Jersey

Phase 4:

* Stage III or IV cancer (per self-report or on the MSKCC EMR). If traditional staging does not apply (i.e. for leukemia), we can allow patient deemed by provider to have poor prognosis/roughly equivalent to Stage III or IV to be referred.
* Age 18 or older
* Of Chinese descent
* Mandarin-speaking
* Have an estimated life expectancy of at least 6 months (per referring physician assessment or on the MSKCC EMR)
* Resides in New York State or New Jersey

Exclusion Criteria:

Phases 1 and 2:

* Presence of cognitive impairment disorder (e.g., delirium or dementia) sufficient to preclude meaningful informed consent and/or data collection. The Chinese version of the Mini Mental State Examination (MMSE) (46) will be used as a cognitive screening tool. Patients with MMSE scores below 20 will be excluded. For English speaking patients we will use the English version of the MMSE.
* Has a household member who has already participated (or agreed to participate).

Phase 3:

* Previous participation in Phases 1 or 2 of the study
* Unable/unwilling to use or no access to a telehealth platform (i.e., telephone or videoconference)
* For participants who express interest in RSMI, unable/unwilling to use Zoom videoconferencing platform
* Unable or unwilling to commit to up to 16 weeks to complete 6-session intervention and follow-up assessments
* Major psychiatric illness or cognitive impairment that in the judgment of study investigators or study staff would preclude study participation
* Patients diagnosed with primary brain tumors (per self-report or on the MSKCC EMR), as they may have difficulty completing the intervention and answering questionnaires
* Undergoing hematopoietic stem cell transplantation (HSCT) (per self-report or on the MSKCC EMR)
* Currently in psychotherapeutic treatment (patients being treated with psychotropic medications will not be excluded, as long as they are not in psychotherapy; per self report)

Phase 4:

* Previous participation in Phases 1, 2, or 3 of the study
* Unable/unwilling to use or no access to the Zoom videoconferencing platform (required for RSMI)
* Unable or unwilling to commit to up to 16 weeks to complete 6-session intervention and follow-up assessments
* Major psychiatric illness or cognitive impairment that in the judgment of study investigators or study staff would preclude study participation
* Patients diagnosed with primary brain tumors (per self-report or on the MSKCC EMR), as they may have difficulty completing the intervention and answering questionnaires
* Undergoing hematopoietic stem cell transplantation (HSCT) (per self-report or on the MSKCC EMR)
* Currently in psychotherapeutic treatment (patients being treated with psychotropic medications will not be excluded, as long as they are not in psychotherapy; per self report)

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Phase I participants will be recruited through MSKCC and referrals provided by Qcc, CCHC, ACS Asian Initiatives, CBWCHC, NYHQ and NYCAAMH and the Cheung and Kan Medical Group.
  Phase 3 and 4 participants will be recruited through MSKCC and referrals provided by community clinicians/collaborating partners. Flyers (Phase 3, Appendix H) in Chinese announcing the study will be distributed through MSKCC and community organizations and hospitals (e.g., QCC, WCMC, NYP LMH, CCHC, ACS Asian Initiatives, CBWCHC, NYHQ, the Cheung and Kan Medical Group and NYCAAMH).
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2027-02-15 (Estimated); Study Completion 2027-02-15 (Estimated)

PRIMARY OUTCOMES:
adapt the Individual Meaning-Centered Psychotherapy (IMCP) | 2 years
  through formative research, including in-depth interviews, to be culturally and linguistically tailored for Chinese immigrant cancer patients (IMCP-Ch), using the Ecological Validity Model (EVM) of Bernal et al. (3) and the Cultural Adaptation Process (CAP) model of Domenech-Rodriquez and Weiling (1). This addresses existential issues using didactics and experiential exercises and has demonstrated efficacy in reducing existential suffering and improving psychosocial functioning among advanced cancer patients.

CONTACTS AND LOCATIONS:
Overall Officials: Florence Lui, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (9):
- United States (9):
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center Suffolk- Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - City College of New York (Data Collection AND Data Analysis), New York, New York
  - MSK at Ralph Lauren (Limited Protocol Activities), New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Uniondale, New York

REFERENCES:
- [Derived] Lui F, Gany F, Espinosa A, Riobo C, Chang F, Narang B, Rodriguez A, Gonzalez J, Niu Y, Chen RY, Jiang R, Leng J. INTERPRETing to increase access to PSYcho-oncology care (INTERPRET-PSY) for cancer patients with limited English proficiency: study protocol for a pilot randomized controlled trial. Pilot Feasibility Stud. 2026 Jan 29. doi: 10.1186/s40814-026-01770-5. Online ahead of print. PMID 41612461
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/